CLINICAL TRIAL: NCT03912714
Title: The Effect of Appendectomy in Ulcerative Colitis Patients With Active Disease: COlonic Salvage by Therapeutic Appendectomy
Brief Title: COlonic Salvage by Therapeutic Appendectomy.
Acronym: COSTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: University Hospital Birmingham (Other)
Responsible Party: Principal Investigator, Willem A. Bemelman, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018_058
Record Dates: First submitted 2018-08-27; First posted 2019-04-11 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Colitis, Ulcerative
Keywords: Appendectomy, Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Laparoscopic appendectomy (Experimental): Laparoscopic appendectomy in therapy refractory ulcerative colitis patients after pre-operative endoscopic biopsies of the appendix
  Interventions: Procedure: Laparoscopic appendectomy; Procedure: Endoscopic appendix biopsies
- Non-active UC (Active Comparator): Patients with non-active ulcerative colitis planned for surveillance colonoscopy will have additional endoscopic appendix biopsies to evaluate the histological characteristics of the appendix.
  Interventions: Procedure: Endoscopic appendix biopsies
- Healthy control (Active Comparator): 'Healthy control' patients (i.e. patients planned for colonoscopy for polyps) will have additional endoscopic appendix biopsies to evaluate the histological characteristics of the appendix.
  Interventions: Procedure: Endoscopic appendix biopsies
- JAK-inhibitor (Active Comparator): JAK-inhibitor in therapy-refractory ulcerative colitis patients
  Interventions: Procedure: Endoscopic appendix biopsies

INTERVENTIONS:
Procedure: Laparoscopic appendectomy — Surgery will be performed under general anaesthesia. The laparoscopic appendectomy can be performed with the use of 3 trocars; one subumbilical, one suprapubic and one in the lower right quadrant of the abdomen. The appendix is removed using a laparoscopic endostapler enabling a safe and complete appendectomy with the cross stapling line at coecal base. Laparoscopic appendectomy will be performed by a gastrointestinal surgeon with sufficient experience in laparoscopic appendectomies (>20).
  Arms: Laparoscopic appendectomy
Procedure: Endoscopic appendix biopsies — Appendix biopsies will only be taken when the scope easily slides into the lumen of the appendix (the scope will not be pushed into the appendix lumen)

SUMMARY:
Rationale: The annual incidence of ulcerative colitis (UC) amounts to 6-8 new cases per 100.000. Patients are initially treated medically, and colitis refractory to medical management is treated surgically, mostly by means of an (emergency) colectomy or a procto-colectomy with ileal J-pouch anastomosis. Over the past 10 years evidence has been accumulating indicating that the appendix has an immunomodulatory role in patients with UC reducing the need for medication and perhaps even colectomy.

Objective: The objective of this prospective observational cohort study is to evaluate the effect of appendectomy on the disease course of patients with active ulcerative colitis despite standard step-up treatment including biologicals compared to usual care. The second objective is to evaluate if it is possible to predict response to appendectomy based on preoperative radiological or endoscopic findings by comparing results to histological characteristics in the resection specimen.

Study design: The design of the study is a multicentre prospective cohort study including patients with active UC despite standard step-up treatment including optimized biological treatment. Patients failing standard step-up medical treatment (including biologicals), that are discussed in the multidisciplinary meeting to be counselled for a JAK-inhibitor (e.g. tofacitinib, filgotinib) or restorative proctcolectomy with ileal-j pouch anastomosis, will be counselled for appendectomy as an alternative treatment option. All patients will undergo colonoscopy before the start of a new treatment according to current guidelines. Biopsies will be taken to histologically confirm ongoing inflammation. Cecal biopsies will be used to correlate histological findings to response to appendectomy. Patients will undergo assessment of the appendix by ultrasound before surgery. All patients will be followed according to study protocol.

Study population: All patients of 16 years and older, with established diagnosis of UC and ongoing disease activity despite standard step-up treatment including optimized biological treatment that are counselled for medication switch to a small molecule JAK-inhibitor or colectomy, will also be counselled for experimental appendectomy. Patients not interested in appendectomy will be asked for consent to collect data according to study protocol and represent the control group.

Group size calculations are based on an improvement in remission rates from 17% in the second line medical group to 40% in the appendectomy group. With a power of 80%, a 2-sided alpha of 0.05, and accounting for 10% loss to follow-up, a total of 67 patients are required in each group.

Intervention: A laparoscopic appendectomy will be performed in day care setting using a laparoscopic endostapler including the cecal base.

Comparison: Usual care consists of small molecule JAK-inhibitor (e.g. tofacitinib, filgotinib) or surgical treatment by restorative proctocolectomy with ileal J-pouch anastomosis.

Main study parameters/objectives: The primary outcome parameter is the number of patients achieving remission (Total Mayo score ≤2) 12 months after appendectomy. Secondary endpoints are reduction of medical therapy, the disease activity as measured with the Mayo score, colectomy rate, the health related quality of life and costs (EQ-5D, EORTC-QLQ-C30-QL and IBDQ), and histological appendix characteristics predictive of response.

DETAILED DESCRIPTION:
The study is designed as a prospective observational cohort study including patients with active ulcerative colitis despite standard step-up treatment including optimized biological therapy. Sixty-seven consecutive patients who are refractory to medical treatment will be recruited to evaluate the effect of the appendectomy on the disease course. Patients not interested in appendectomy will be asked for consent to collect all data according to study protocol and represent the control group. These patients either receive switch in medical treatment to the small molecule JAK-inhibitor (e.g. tofacitinib, filgotinib or upadacitinib) or a procto-colectomy.

All eligible patients will be extensively counselled about these three treatment options at the outpatient clinics by a gastroenterologist and/or surgeon. Patients who failed small molecules can be counselled for appendectomy if not done so when initially counselled for treatment with small molecules. Patients with presumed therapy-refractory inflammation will undergo ileocolonoscopy, which is part of standard daily practice. Active disease is required for inclusion, and is defined as a combined clinical and endoscopic Mayo-score of ≥5 with an endoscopic subscore of 2 or 3. Patients will also undergo preoperative ultrasound to assess clinical characteristics of the appendix preoperatively.

After inclusion, a laparoscopic appendectomy will be performed within 9 weeks. Patients will be followed 3, 6, 12 and 30 months after laparoscopic appendectomy to assess the patients' clinical condition and the non-invasive Mayo score. According to standard practice evaluating therapy change, an endoscopy including biopsies of colon and cecal base 12 months after appendectomy will be performed to assess mucosal appearance and complete the Mayo score.

Postoperatively, patients will receive the similar medical treatment as given pre-appendectomy. If medication can be tapered post-appendectomy, this will be done according to the experience of the treating physician and current guidelines. Patients will complete health related quality of life questionnaires (EQ-5D, EORTC-QLQ-C30-QL and IBDQ) at inclusion and at 3, 6, 12 and 30 months follow-up, alongside the MYMOP at inclusion and 12 months follow up via email or a telemedicine application (MyIBDcoach).

The preoperative ultrasound findings and endoscopic cecal biopsies will be used to analyse if histological inflammation in the appendix resection specimens can be reliably predicted. Histological findings in the resection specimens will be correlated to clinical and pathological response after appendectomy. Furthermore, in 20 patients who are planned for colonoscopy (10 patients with non-active UC and 10 non-UC patients with polyps) additional cecal biopsies will be taken to use as a reference control group

ELIGIBILITY:
Inclusion criteria (study group)

* Age 16 years and older
* Established diagnosis of UC
* Active disease (defined both clinically and endoscopically as Mayo-score ≥5 with endoscopy score of 2 or 3) despite standard step-up treatment including biological treatment
* Obtained written informed consent

Inclusion criteria (control group)

* Age 16 years and older
* UC patients with non-active disease (defined both clinically and endoscopically as Mayo-score ≤5 with endoscopy score of 0 or 1) or non-UC patients with polyps
* Planned colonoscopy
* Obtained written informed consent

Exclusion criteria (study group)

* Prior appendectomy or other abdominal surgery by laparotomy precluding safe appendectomy
* Suspicion of Crohn's disease.
* Toxic megacolon or severe acute colitis necessitating clinical admission.
* History or suspicion of colonic dysplasia or malignancy.
* Required daily oral prednisone dose exceeding 20 milligrams.
* Patients with active extra-intestinal infections, liver or kidney failure, mayor lung and heart co-morbidity.
* Insufficient command of Dutch or cognitively unable to complete Dutch questionnaires.

Exclusion criteria (histological control group)

* Prior appendectomy.
* Suspicion of Crohn's disease.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Remission rate | 12 months
  Steroid-free remission rate (Total Mayo Score ≤2, with no individual sub-score exceeding 1 point) 12 months after appendectomy without switch of therapy.

SECONDARY OUTCOMES:
Reduction of medical therapy including corticosteroids | Every 3 months, up to 12 months
  Downscaling of medical therapy including corticosteroids (number of patients that stop medication).
Disease activity, as measured with the full Mayo score | 6 and 12 months
  Using this 12-point scoring system, disease activity is evaluated based on stool frequency, rectal bleeding, the physician's global assessment, and endoscopic appearance. Each subscale is ranging from 0-3 and higher values represent worse outcomes. The full Mayo score is computed by the sum of the four subscores.
Failure | Every 3 months, up to 12 months
  Defined as colectomy, switch of biological treatment, (re)start of corticosteroids or start of trial medication after a minimum of 1 month postoperative.
Health related quality of life (EQ-5D) | 3, 6 and 12 months
  This questionnaire is a simple, generic instrument for describing and valuing health related quality of life. It includes 5 items (mobility, personal care, daily activities, pain, and anxiety/ depression) that are answered on a 3-point scale ranging from no problems (level 1) to extreme problems (level 3).
Disease specific quality of life (IBDQ) | 3, 6 and 12 months
  A disease-specific questionnaire that measures quality of life in 4 domains (bowel symptoms, systemic symptoms, social function, and emotional function). The IBDQ consists of 32 questions which are rated on a scale from 1 to 7, resulting in a total score ranging from 32 to 224 and a higher score represents a better quality of life.
Time to remission | Every 3 months, up to 12 months
  Time between inclusion and remission
Pathological analysis of resection specimen to determine histological characteristics according to the Geboes score, predictive of response . | Baseline
  Geboes score less than 3: (grade 0-5: architectural changes, increase of chronic inflammatory infiltrate, increase of eosinophils in the lamina propria, increase of neutrophils in the lamina propria, involvement of neutrophils in the epithelium (cryptitis), crypt destruction, and erosion or ulcerations)
Global quality of life (EORTC-QLQ-C30-QL) | 3, 6 and 12 months
  This sub questionnaire contains the 2 items of the global quality of life dimension of the EORTC-QLQ-C30 questionnaire. It includes 30 questions, and answers are ranging from no problems (1 point) to extreme problems (4 points).

CONTACTS AND LOCATIONS:
Overall Officials: Christianne Buskens, MD, PhD, Principal Investigator — Amsterdam Medical Centre
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Visser E, Reijntjes MA, Heuthorst L, Stellingwerf ME, West R, van Dongen K, Crolla RMPH, van Dieren S, van der Bilt JDW, Bemelman WA, D'Haens GR, Buskens CJ; COSTA Study Group. Appendicectomy versus switching to a JAK inhibitor in inducing remission in patients with active ulcerative colitis after biologic therapy failure (COSTA): 1-year results of a multicentre, prospective, cohort study. Lancet Gastroenterol Hepatol. 2026 Jan 6:S2468-1253(25)00291-2. doi: 10.1016/S2468-1253(25)00291-2. Online ahead of print. PMID 41512889